CLINICAL TRIAL: NCT04072276
Title: Long-Term Immunogenicity Study of Inactivated EV71 Vaccine Produced in Vero Cells With Adjuvant AlPO4 in Children: Extension Study of Protocol CT-EV-21
Brief Title: Long-Term Immunogenicity Study of Inactivated EV71 Vaccine in Children
Status: Completed | Type: Observational
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: FU-EV-21e
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2021-09

CONDITIONS: Enterovirus 71 Human
Keywords: EV71 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EV71 Vaccine with Adjuvant AlPO4: EV71 Vaccine Produced in Vero Cells with Adjuvant AlPO4
  Interventions: Biological: EV71 vaccine
- Adjuvant AlPO4: Placebo (Adjuvant AlPO4 only)
  Interventions: Biological: EV71 vaccine

INTERVENTIONS:
Biological: EV71 vaccine — EV71 vaccine with Adjuvant AlPO4 and the placebo (Adjuvant AlPO4 only) were randomly administrated to subject in CT-EV-21 study

SUMMARY:
This study is designed to evaluate the long-term antibody titers of EV71 vaccine 4 and 5 years after first dose vaccination for subjects at the age of 2 to < 6 years , and 3 to 5 years after first dose vaccination for subjects at the age of 2 months to < 2 years

DETAILED DESCRIPTION:
This is an extension study of protocol CT-EV-21, to evaluate the long-term immunogenicity of EV71vaccine.

The first study visit will be approximately 3 or 4 years after the administration of first vaccination of EV71 vaccine or placebo in CT-EV-21 study; 4 years after the first vaccination for subjects 2 to < 6 years of age (2b), and 3 years after first dose for subjects 2 months to < 2 years of age (2c and 2d).

Subjects of 2b will remain in the study for approximately 12 months and will have 2 clinic visits; subjects of 2c and 2d will remain in the study for approximately 24 months and will have 3 clinic visits. Immunogenicity response against EV71 virus antigen at each visit will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed participation in study CT-EV-21 part 2b, 2c, and 2d, and have received protocol specified doses of EV71 vaccine or Placebo (total of 2 doses in part 2b, and 3 doses for part 2c and 2d).
* The subjects' guardians are able to understand and sign the informed consent form.

Exclusion Criteria:

* Subjects and/or guardians who refuse to comply with the study procedures

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects who have completed participation in study CT-EV-21
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Serum neutralizing antibody titer | Up to 5 years after first dose of EV71 vaccination
  Geometric mean titer (GMT) of EV71 neutralizing antibody titers at 4 and 5 years after first dose of EV71 vaccination for subjects of 2b; and 3 to 5 years after first dose of EV71 vaccination for subjects of 2c and 2d.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital; Cheng-Hsun Chiu, M.D., Ph.D., Principal Investigator — Chang Gang Memorial Hospital, LinKou; Chien-Yu Lin, M.D., Ph.D., Principal Investigator — Mackay Memorial Hospital, HsinChu; Nan-Chang Chiu, M.D., Principal Investigator — Mackay Memorial Hospital
Locations (4):
- Taiwan (4):
  - Mackay Memorial Hospital, HsincChu, Hsinchu
  - Mackay Memorial Hospital, Taipei, Taipei
  - National Taiwan University Hosptial, Taipei
  - Chang Gung Memorial Hospital, LinKou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No